CLINICAL TRIAL: NCT04745494
Title: Studies of Mothers With Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16/0679
Record Dates: First submitted 2020-03-25; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Postnatal Depression
Keywords: Oxytocin
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, case-controlled, randomised controlled-trial, within-subjects, cross-over design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT administration (Active Comparator): All participants will receive a single dose of 24IU OT (40.32µg, Syntocinon) delivered via a nasal spray.
  Interventions: Other: OT administration
- Placebo administration (Placebo Comparator): All participants will receive a single dose of a placebo delivered via a nasal spray.
  Interventions: Other: Placebo administration

INTERVENTIONS:
Other: OT administration — OT nasal administration
  Arms: OT administration
Other: Placebo administration — Placebo nasal administration
  Arms: Placebo administration

SUMMARY:
This study investigates the effects of a single dose of oxytocin (OT) delivered via a nasal spray in women with and without traits of postnatal depression (PND).

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, case-controlled, randomised controlled-trial, within-subjects, cross-over design will be conducted.

Participants will include mothers and their infant in the postnatal period. All participants will be screened for symptoms of low mood on the Edinburgh Postnatal Depression Scale (EPDS) and then assigned into 2 groups comprising probable PND cases and controls.

All participants will take part in 3 conditions at Baseline (before nasal spray administration), Condition 1 (after first OT/Placebo administration) and Condition 2 (after second OT/Placebo administration), and will complete the same order of tasks.

ELIGIBILITY:
Inclusion Criteria:

* All mothers will be aged ≥18 years old.
* Mothers in the clinical group will score above the clinical cut-off point on the EPDS.
* Mothers in the control group will score below the clinical cut-off point on the EPDS.
* Mothers must be able to read and write English at a level sufficient to complete study related assessments.

Exclusion Criteria:

* If the mother is younger than 18 or post-menopausal
* If the pregnancy was a result of fertility treatment
* If the mother is pregnant
* If the mother has history of psychotic illness
* If the mother is at risk of self-harm
* If the mother is involved in other active drug trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change in maternal mood | Baseline, 35-45 minutes after intervention administration
  Change in maternal mood will be assessed using the PANAS questionnaire

SECONDARY OUTCOMES:
Change in maternal mindmindedness | Baseline, 35-45 minutes after intervention administration
  Change in maternal mindmindedness will be assessed using Meins' Mindmindedness Manual
Change in mother-infant interactional style | Baseline, 35-45 minutes after intervention administration
  Change in mother-infant interactional style will be coded using Feldman's Coding Interactive Behaviour Manual
Change in maternal OT | Baseline, 35-45 minutes after intervention administration
  Change in maternal salivary and breast milk OT will be assayed
Change in infant OT | Baseline, 35-45 minutes after intervention administration
  Change in infant salivary OT will be assayed
Maternal gaze during interaction with her infant | 35-45 minutes after intervention administration
  Maternal gaze will be assessed using a Tobii X2-30 eye tracker

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, UK, United Kingdom

REFERENCES:
- [Derived] Lindley Baron-Cohen K, Feldman R, Fearon P, Fonagy P. Intranasal oxytocin administration improves mood in new mothers with moderate low mood but not in mothers with elevated symptoms of postnatal depression: A randomised controlled trial. J Affect Disord. 2022 Mar 1;300:358-365. doi: 10.1016/j.jad.2021.11.062. Epub 2021 Nov 26. PMID 34843839